CLINICAL TRIAL: NCT02164123
Title: Autonomic Effects of T4 Mobilization in Asymptomatic Subjects: Randomized Clinical Trial
Brief Title: Autonomic Effects of T4 Mobilization in Asymptomatic Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Francisco Xavier de Araujo, Pt, Pt, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UFCSPA-FXA-01
Record Dates: First submitted 2014-06-09; First posted 2014-06-16 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Other Disorders of the Autonomic Nervous System; Vertebra; Degeneration
Keywords: Autonomic effects; spinal mobilization; clinical trial
MeSH Terms: interventions — Prone Position; Sitting Position

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Spinal mobilization (Experimental): 20 subjects will be randomized to this arm. A postero-anterior (PA) mobilization, to the fourth thoracic vertebra will be applied, for 3 sets of one minute. The subject will be comfortable prone lying.
  Interventions: Other: Spinal mobilization
- Spinal Mobilization II (Active Comparator): 20 subjects will be randomized to this arm. A postero-anterior (PA) mobilization, to the fourth thoracic vertebra will be applied, for 3 sets of one minute, but in this case, the subject will be seated, in a position that influence the sympathetic trunk, at the thorax.
  Interventions: Other: Spinal Mobilization II
- Placebo (Placebo Comparator): 20 subjects will be randomized to this arm. Only manual contact will be applied, without any oscillation. The subject will be comfortable prone lying. The intervention time is the same of the other arms.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Spinal mobilization — Experimental group
  Other Names: Postero-anterior spinal mobilization in prone
  Arms: Spinal mobilization
Other: Spinal Mobilization II — Active comparator group
  Other Names: Postero-anterior spinal mobilization in seated position
  Arms: Spinal Mobilization II
Other: Placebo — Placebo group
  Other Names: Placebo technique, olny manual contact
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether passive accessory intervertebral mobilization applied to the fourth thoracic vertebra produces autonomic effects.

DETAILED DESCRIPTION:
Asymptomatic subjects will be recruited to this study. Pressure pain threshold, heart rate, heart rate variability and skin conductance will be measured before, immediately after and fifteen minutes after the intervention.

Subjects will be randomized into three groups: Passive accessory intervertebral mobilization one, passive accessory intervertebral mobilization two and placebo group.

The researcher that will do the intervention will be blinded to the outcomes measures, and the researcher that will do the measurements will be blind to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic subjects
* Aged between 18 - 40 years old
* Portuguese readers and writers

Exclusion Criteria:

* History of lesion or surgery to the spine

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2014-07; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Skin conductance | Change from Baseline imediately after, and 15 minutes after the intervention
  Skin conductance will be measured with Biopac MP150, the electrodes will be attached to the third and fourth fingers bilaterally. This measurement will be made during all the procedure, before, during and until 15 minutes after the intervention.

SECONDARY OUTCOMES:
Pressure pain threshold | Change from Baseline imediately after, and 15 minutes after the intervention
  Pressure pain threshold will be measured with a digital algometer (Model FDX 10; Wagner Instruments, Greenwich, CT). This measurement will be made on the spinous process of C5 and T4, on the first dorsal interossei, and on the anterior tibial tuberosity bilaterally.

OTHER OUTCOMES:
Heart rate variability | Change from Baseline imediately after the intervention
  Heart rate variability will be measured with a Polar Advantage Interface (Polar Electro Oy, Kempele, Finland). The belt will be positioned centrally, directly below the xiphisternum. Heart rate data acquisition will me made for 5 minutes at baseline and for 5 minutes immediately after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco De Araujo, Pt, Principal Investigator — Federal University of Health Science of Porto Alegre
Locations (1):
- Universidade Federal de Ciências da Saúde de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil